CLINICAL TRIAL: NCT01626547
Title: Biosimilar Retacrit™ (Epoetin Zeta) in the Treatment of Chemotherapy-Induced Symptomatic Anaemia in Haematology and Oncology; Non-interventional, Observational, Prospective Study
Brief Title: Biosimilar Retacrit™ (Epoetin Zeta) in the Treatment of Chemotherapy-Induced Symptomatic Anaemia in Haematology and Oncology
Status: Completed | Type: Observational
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: ORHEO
Record Dates: First submitted 2012-06-07; First posted 2012-06-22 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2015-07

CONDITIONS: Chemotherapy-induced Symptomatic Anaemia; Solid Tumours; Malignant Lymphomas; Multiple Myeloma
Keywords: symptomatic anameia
MeSH Terms: conditions — Lymphoma; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to observe correction of haemoglobin (Hb) levels in patients receiving chemotherapy as a consequence of a solid tumour, a malignant lymphoma or a multiple myeloma and who are treated with Retacrit™.

DETAILED DESCRIPTION:
This is a non-interventional, descriptive, national, multi-site, longitudinal and prospective observational study in adult patients who are suffering from cancer or malignant blood disease and whose chemotherapy treatment has induced symptomatic anaemia and being treated with Retacrit® to correct haemoglobin levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥18 years .
* Patients present with chemotherapy-induced symptomatic anaemia.
* Patients suffer from solid tumours, malignant lymphomas or multiple myeloma and have developed symptomatic anaemia due to their chemotherapy.

  * The patients may be included regardless of their chemotherapy cycle (from the first cycle until the last cycle)
* Patients eligible for epoetin alfa biosimilar treatment.

Exclusion Criteria:

* Patients are not receiving chemotherapy.
* Patients already included in an epoetin zeta study.
* Patients presenting with the contraindications to epoetin zeta.
* Patients presenting with the hypersensitivity to the active substance or any of the excipients.
* The patient presents erythroblastopenia, or 'pure red cell aplasia' (PRCA).
* Patients with uncontrolled hypertension.
* Patients who cannot receive adequate prophylaxis by antithrombotic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chemotherapy-induced symptomatic anaemia. Patients suffer from solid tumours, malignant lymphomas or multiple myeloma and have developed symptomatic anaemia due to their chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change and corrected Hemoglobin levels | 6 months
  Participants who have hemoglobin values between 11 and 12 g/dl after 6 months of treatment.

SECONDARY OUTCOMES:
Observation of blood value development | 6 months
  Observation of blood value development: hemoglobin, hematocrit, reticulocytes, serum iron, ferritin, transferrin saturation
Evaluation of the profiles of treated patients | 6 months
Evaluation of prescriber's therapy plan | 6 months
Evaluation of the correlation between the therapy plans of prescribing oncologists and patient characteristics | 6 months
Observation of the tolerability profile of Epoetin Zeta | 6 months

CONTACTS AND LOCATIONS:
Locations (34):
- Germany (34):
  - Alzey
  - Bad Säckigen
  - Berlin
  - Bonn
  - Borken
  - Brandenburg
  - Chemnitz
  - Cottbus
  - Essen
  - Frankenthal
  - Garbsen
  - Halberstadt
  - Hanover
  - Herne
  - Holzkirchen
  - Krefeld
  - München
  - Münster
  - Neuss
  - Nuremberg
  - Oberhausen
  - Olpe
  - Oranienburg
  - Paderborn
  - Parchim
  - Plauen
  - Remscheid
  - Rodgau
  - Rötha
  - Schönebeck
  - Soest
  - Stralsund
  - Stuttgart
  - Velbert